#### 1. Hypothesis and Specific Aims

Overarching Hypothesis: Insulin signaling is a critical neurobiological substrate of anhedonia in mood disorders

<u>Specific Hypotheses:</u> In individuals with mood disorders, objective and self-reported measures of anhedonia and reward behaviors are associated with alterations in insulin signaling-related molecular, cellular and neural substrates. Considering the role of insulin in the regulation of energy expenditure, we primarily hypothesize that individuals with mood disorders will display decreased willingness to make effort for rewards, relative to healthy controls; and that this abnormality will be associated with:

- a) Molecular: Differential gene and protein expression of the metabolic (i.e. PI3K/Akt) and mitogenic (i.e. Ras/MAP kinase) components of the insulin signaling pathway, as well as with components of reward-related processes (i.e. dopamine receptors and transporter)
- b) Physiology: Reduced peripheral sensitivity to insulin and corresponding metabolic correlates, including increased body mass index and dyslipidemia (i.e. peripheral insulin resistance)
- c) Neural Circuits: Diminished response to insulin in cortico-striatal networks (i.e. brain insulin resistance)

Overarching Aim: To determine the role of insulin signaling on the neurobiological substrates subserving anhedonia within individuals with mood disorders.

## Specific Aims:

- a) Molecular: Assessment of components of the insulin cascade, as well as of anhedonia and reward-related processes, using a proteomics and gene expression approach;
- b) Physiology: Measurement of peripheral sensitivity to insulin and metabolic correlates, including body mass index and dyslipidemia;
- c) Neural Circuits: Evaluation of the insulin sensitivity of prefrontal (e.g. prefrontal cortex) and striatal (e.g. nucleus accumbens, ventral tegmental area) networks in the resting-state and during an effort-based decision making test, using acutely administered intranasal insulin and functional magnetic resonance imaging (fMRI);
- d) Behavioral: Measurement of willingness to make effort for rewards, as well as of other components of reward response and anhedonia, using validated behavioral tasks and clinical scales (e.g. Snaith-Hamilton Pleasure Scale SHPS).

#### 2. Background and Rationale

Mood disorders (i.e. major depressive disorder [MDD] and bipolar disorder [BD]) and metabolic disorders (i.e. type 2 diabetes mellitus [T2DM], obesity) are highly prevalent and impactful conditions. Epidemiological studies have identified depressive disorders and diabetes as leading causes of disability worldwide<sup>1</sup>. Mood and metabolic disorders are also major causes of excessive and premature mortality. Mortality studies indicate that with individuals with MDD or BD have markedly reduced life expectation, on average of 10-15 years<sup>2</sup>; the main driver of excess and premature mortality in this population is cardiovascular disease and/or diabetes complications<sup>2,3</sup>. Conversely, depressive symptoms, particularly anhedonia, are consistently reported in T2DM populations and have been associated with an increased incidence of complications and all-cause mortality<sup>4,5</sup>.

Comorbid metabolic disorders are extremely common in individuals with mood disorders. Metaanalytic studies have documented that individuals with MDD or BD have an approximately 2-fold increased risk of T2DM, relative to the general population<sup>6</sup>. It is estimated that the prevalence of

T2DM in individuals with mood disorders is between 8 and 10%, whereas the prevalence of metabolic syndrome is approximately 30%<sup>7</sup>. Convergent lines of inquiry indicate that mood and metabolic disorders have a bidirectional association<sup>8-10</sup>. For example, it is reported that individuals with T2DM have an approximate 2-3 fold greater risk for subsequently declaring MDD or BD<sup>11</sup>. Nonetheless, the association between metabolic and mood disorders is still poorly understood. Overlapping risk factors (e.g. diet, physical activity, psychotropic medications, sleep, childhood trauma) have an important role<sup>6</sup>; however there is insufficient data on the extent to which these environmental factors are responsible for the mood-metabolic disorders comorbidity. Mechanistic studies have documented a role for the biological substrates of metabolic and mental disorders, such as neurostructural alterations <sup>12,13</sup>, and differences in peripheral biomarkers<sup>14</sup>. A recent genetic study identified multiple genes that are likely shared between mood and metabolic disorders; pathway analysis revealed an over-representation of genes that encode for molecules involved in dopamine signaling<sup>15</sup>. There is considerable evidence that dopamine has a core role in anhedonia and reward-related behaviors, indicating that this is a particularly promising area for further advancing the knowledge on the association of mood and metabolic disorders.

#### 1.1. Mood Disorders and Anhedonia

Anhedonia is defined as markedly diminished interests or pleasure in all, or almost all, activities most of the day, nearly every day for an extended period of time. Anhedonia is a core criterion item for the diagnosis of a major depressive episode. Anhedonia is also a robust predictor of poorer longitudinal course of symptoms of MDD and BD<sup>16-19</sup>. Existing psychological and pharmacological treatments are relatively ineffective for treating anhedonia, as standard medication treatments have little effect and in some cases may even worsen anhedonic symptoms<sup>17,20</sup>. As a result, anhedonia has been described as one of the most prevalent residual disturbances following treatment with selective serotonin re-uptake inhibitors 17,21,22.

Anhedonia includes elements of multiple reward processes<sup>23-25</sup>. Reward systems are primarily responsible for responses to positive motivational situations or contexts, such as reward seeking, and reward/habit learning<sup>23-25</sup>. Reward is a broad and heterogeneous construct. To effectively study it, it is important to consider its three main subconstructs: (1) reward responsiveness, including anticipatory and initial hedonic responses; (2) learning, or the acquisition of information about stimuli, actions and context; and (3) valuation, including the measurement of value and/or incentive salience of a prospective outcome and the willingness to work for it (i.e. effort)<sup>26,27</sup>.

Evidence indicates that individuals with mood disorders exhibit abnormalities in multiple of these reward subcomponents<sup>28-32</sup>. Anhedonia is closely related to reward anticipation, motivation and decision making<sup>29,33</sup>. A consistent finding has been a decrease in the willingness to expend effort and/or in the modulation of effort expenditure for rewards<sup>28-31,33</sup>. It has been demonstrated that individuals with depression display reduced motivation on effort-based decision making<sup>29-31</sup>, a dissociation between liking a reward and the willingness to exert effort for it<sup>28</sup>, an increased subjective feeling of having exerted more effort<sup>31</sup> and a lower ability to effectively use information about rewards to modify their behavioral choices<sup>29</sup>.

#### 1.2. Neural Substrates of Anhedonia and Reward

The most well-characterized reward circuit is the mesolimbic pathway, which consists of dopaminergic projections from the ventral tegmental area (VTA) to the nucleus accumbens (NAc)<sup>34,35</sup>. These areas are heavily interconnected with the prefrontal cortex (PFC), amygdala and hippocampus, among other areas<sup>34</sup>. Specifically, connections between the dorsolateral PFC (dlPFC), NAc and VTA

have a key role in motivated behavior<sup>36</sup>. Indeed, connectivity between the PFC and striatal areas during reward-related tasks negatively correlates with anhedonia in individuals with MDD<sup>37,38</sup>.

Dopaminergic neurotransmission has been highlighted as a key component of multiple reward processes<sup>39</sup>. Dopamine signaling has traditionally been implicated in arousal, motivation and psychomotor activation (i.e. incentive salience models), and reward learning/reinforcement (i.e. prediction error models)<sup>40-42</sup>. Recent work proposes that dopamine signals value, or the available reward for a certain effort, which is then employed for both learning and motivational functions<sup>42</sup>. Multiple studies from different lines of research, such as genetics, neuroimaging and pharmacology, have documented abnormalities in dopaminergic neurotransmission in individuals with mood disorders (8, 9). For example, neuroimaging studies have demonstrated alterations in dopamine receptor and transporter binding in individuals with MDD<sup>43-45</sup>. Conversely, the Val(158)Met polymorphism of the catechol-O-methyltransferase (COMT) gene, which affects dopamine catabolism and modulates prefrontal dopamine levels, has been associated with measures of anhedonia<sup>46,47</sup>. Overall, abnormalities in reward-related behaviors and dopaminergic transmission are well-established features of mood disorders phenomenology and neurobiology.

#### 1.3. Brain Insulin Signaling Pathway, Dopamine Signaling and Reward

Dopamine signaling within and across brain circuits is in interplay with many systems relevant to reward, including the insulin signaling pathway<sup>34,48,49</sup>. Insulin acts via the insulin receptor (INSR). Activation of INSR initiates the recruitment of the insulin receptor substrate (IRS) family of proteins, which organize and mediate signaling cascades<sup>50,51</sup>. IRS1 and IRS2 are the most extensively studied substrates; they are expressed in the brain and have well-documented effects on insulin signaling and glucose homeostasis<sup>52-54</sup>. Insulin binding to INSRs activates several divergent signaling pathways, including the metabolic pathway (i.e. PI3K/Akt), which affects glucose and lipids homeostasis; and the mitogenic pathway (i.e. Ras/MAP kinase), which is implicated in the regulation of apoptosis and cell proliferation/differentiation.

Multiple brain regions that are relevant to reward systems have relatively increased expression of INSRs (e.g., PFC, hippocampus, amygdala, substantia nigra)<sup>22,23</sup>. Specifically, midbrain dopamine neurons widely express INSRs<sup>49</sup>. Imaging studies have reported that, in healthy individuals, insulin modulates brain activity in the hypothalamus, hippocampus and prefrontal cortex<sup>34-36</sup>. Brain insulin signaling has traditionally been implicated in glucose and lipid metabolism, and eating behavior. However, replicated evidence, from multiple studies, has documented that insulin also has a role on emotional processing<sup>55-57</sup> and reward processes, including, but not limited to, those pertaining feeding behaviors and energy expenditure<sup>58,59</sup>.

An important way insulin affect reward processes is via interaction with dopaminergic signaling. Evidence indicated that insulin modulates multiple components of dopamine transmission, including synthesis and transport, receptors function and reuptake and degradation. For example, lower expression and function of tyrosine hydroxylase (TH), the rate-limiting enzyme in dopamine biosynthesis, have been reported in animal models of diabetes<sup>60,61</sup>. In humans, insulin resistance was associated with less endogenous dopamine at D2/3 receptors in the ventral striatum and NAc, in both obese and non-obese participants<sup>62,63</sup>. A separate study documented that weight loss following bariatric surgery was associated with an increase in D2 receptor availability<sup>64</sup>.

Termination of dopamine action, which is via reuptake from the synaptic cleft by the dopamine transporter (DAT), or by degradation by monoamine oxidases (MAOs) A/B and COMT, has also been shown to be affected by insulin. Studies with animal models of diabetes have reported lower availability and activity of DAT<sup>65,66</sup> and lower activity of COMT<sup>67</sup>; whereas a murine model with a

brain specific knockout of the insulin receptor reported that decreased insulin function in the brain resulted in increased expression of MAO A/B in the striatum and NAc<sup>68</sup>. As a result, evidence indicates that insulin sensitivity modulates reward behavior in obese adults, wherein insulin resistance was associated with a stronger preference for immediately receiving a smaller, but certain, monetary reward over delaying the receipt of a larger, but less certain one (i.e. greater delay discounting)<sup>69</sup>.

# 1.4. Insulin Signaling, Anhedonia and Major Depressive Disorder

The epidemiological, phenomenological and biological associations between mood disorders and metabolic disturbances have been amply documented. The foregoing observations provide the rationale for hypothesizing that there is a neurobiological association between metabolic disorders (e.g. diabetes) and mood disorders. The devastating impact of mood and metabolic disorders on affected individuals underscores the importance of urgently understanding better the basis of this association. Anhedonia is a well-described symptom that similarly occurs in both disorders. The extant evidence of the association between insulin and dopamine signaling and the potential repercussions of disturbances in this system indicates that this is a promising target for clinical and neurobiological investigations. The interface between anhedonia and insulin represents a unique opportunity to integrate innovative and transdisciplinary lines of research in an investigative platform aiming at providing a more accurate and refined assessment of relevant mechanisms in the mood-metabolic disorders comorbidity.

## 2. Preliminary Data

Using the "Gene Expression in Postmortem DLPFC and Hippocampus from Schizophrenia and Mood Disorders" (dbGaP accession number phs000979.v1.p1) database, which contains microarray data from the post-mortem dlPFC (healthy controls [HC]: n = 209; patients: n = 321) and hippocampus (HC: n = 180; patients: n = 196), we conducted a hypothesis-driven analysis through the a priori selection of 12 dopamine- and 3 insulin-related genes (manuscript under review). Results showed that, in the dlPFC, after adjustment for relevant covariates, expressions of insulin receptors- (i.e. INSR, IRS1/2) and dopamine regulation-related genes (e.g. TH, DRD1-5, DAT) were influenced by body mass index (BMI), with significantly lower expression in high BMI patients with mood or psychotic disorders (Figure 1). In the hippocampus, we observed significantly lower expressions of these genes, which were not affected by BMI.

Genes that were differentially expressed between groups were selected for mediation analyses. Diagnosis by BMI effects on expression of dopamine genes were fully mediated by expression of INSR. Analysis of conditional indirect effects showed interactions between INSR and BMI, indicating significantly stronger indirect effects at higher BMI values. In the hippocampus, we observed that expression of insulin receptor substrate 1 and 2 fully mediated the effects of diagnosis on expression of dopamine genes (Figure 2). All models were significant (e.g. DRD1:  $R^2 = 0.31$ ,  $F_{6,385} = 29.519$ , p < 0.001). These results suggest that the differential expression of dopamine-related molecules in the postmortem brain of individuals with mental disorders is related to altered expression of insulin signaling genes. We also observed that obesity has region-specific moderating effects on gene expression and co-expression, supporting the hypothesis that metabolic systems are critical mediators of dopaminergic function and providing the rationale for further investigation.

Figure 1 – Mean standardized expression values of insulin and dopamine signaling genes in the dorsolateral prefrontal cortex, according to group (HC vs. MI) and obesity (BMI  $\geq$  30 kg/m<sup>2</sup>). HC: healthy controls; MI: mental illness; BMI: body mass index.



Figure 2 – Unstandardized path coefficients for a mediation model in the hippocampus, adjusted for age, gender, race, ethanol and nicotine/cotinine. \* p < 0.05; \*\* p < 0.001.



Rodrigo B. Mansur Research Proposal Project Title: Anhedonia and the insulin pathway: a mechanistic nexus for the mood and metabolic disorders comorbidity

## 3. Design and Methodology

<u>Study population:</u> We propose to recruit 50 adults between the ages of 18 to 50 years: 25 patients with DSM-5 defined MDD or BDI/II, in a depressive episode, recruited from the Mood Disorder Psychopharmacology Unit, University Health Network, and 25 age- and sex-matched healthy controls recruited through local advertisements in the community.

# <u>Inclusion criteria (patients):</u>

- 1. Age 18-50
- 2. DSM-5 defined MDD/BD and a total score ≥20 on the Montgomery-Åsberg Depression Rating Scale (MADRS) and no history of dementia or intellectual disability
- 3. A written, voluntary informed consent prior to study enrollment

# Exclusion criteria (patients):

- 1. Use of insulin and/or oral hypoglycemiants, due to its confounding effects
- 2. Diagnosis of possible or probable AD, MCI, or any other dementia
- 3. History of neurological disorder, or evidence of neurologic or other physical illness that could produce cognitive deterioration
- 4. Substance use disorder within 3 months before screening or a positive baseline toxicology screen
- 5. Presence of clinically unstable general medical illness
- 6. Pregnancy or breastfeeding
- 7. MRI contraindications

# <u>Inclusion criteria (healthy controls):</u>

- 1. Age 18-50
- 2. A written, voluntary informed consent prior to study enrollment

#### Exclusion criteria (healthy controls):

- 1. Use of insulin and/or oral hypoglycemiants, due to its confounding effects
- 2. Presence of any current or lifetime psychiatric or neurological conditions
- 3. Substance use disorder within 3 months before screening or a positive baseline toxicology screen
- 4. Presence of clinically unstable general medical illness
- 5. Pregnancy or breastfeeding
- 6. MRI contraindications

<u>Study Procedures:</u> Single-dose, randomized, controlled, double-blinded, cross-over study (50 participants)

Screening and Baseline Assessment: Patients and healthy controls will first meet, in-person or virtually, with a staff psychiatrist for a clinical consultation or a research team member, respectively. After obtaining consent and if inclusion criteria are met, a medical comorbidity questionnaire will be administered to screen for concurrent and lifetime medical conditions. Participant's demographic characteristics and current medications, as well as lifetime psychotropic medications received will be recorded. We will also assess dietary intake with the Diet History Questionnaire III (DHQ III); smoking, by questioning number of cigarettes smoked per day, age when smoking started, and quitting date, if applicable, to calculate a smoking pack-year history; physical activity using the International Physical Activity Questionnaire (IPAQ); and alcohol and/or substance abuse. In addition, we will assess demographics, socioeconomic status, medical history, and family psychiatric history; childhood trauma history with the Childhood Trauma Questionnaire (CTQ) will also be assessed. Participants will also be asked to complete an MRI screening questionnaire to ensure that they have no contraindications. The following self-reported measures will be carried out: Perceived Deficits Questionnaire-Depression (PDQ-D), Sheehan Disability Scale (SDS), UCLA life Stress (Episodic), DeJong Gierveld Loneliness Scale, and Pittsburg Sleep Quality Index (PSQI) (Table 1).

When in-person visits are possible, participants will complete a urine drug screen. Female participants will be asked to do blood work to confirm they are not pregnant.

Physiological Assessment: Anthropometric (i.e. BMI, waist-hip ratio) and metabolic measurements (i.e. fasting glucose, fasting insulin, glycated hemoglobin, lipids and HOMA-IR) will be completed at each study visit (1-3). In addition, physical activity and energy expenditure will be measured using an accelerometer. Participants must wear the accelerometer at all times for one week and return it upon Visit 3 for data collection and analysis. Additionally, a heart rate monitor device will be connected to the accelerometer that will monitor heart rate variability over one day of the week that the subjects wear the accelerometer.

Laboratory Assessment:

**Routine**: the following laboratory tests will be completed:

| Triglycerides |
|--------------------|
| Total Cholesterol |
| Insulin |
| Glucose |
| HbA1c |
| C-Peptide |
| IGF-1 |
| TSH |
| Free T4 |
| Free T3 |
| C-Reactive Protein |
| hCG |

**Biomarkers:** High sensitivity CRP and TNF $\alpha$  will be measured at both visits (hs-CRP only). Ultrasensitive ELISA will be used to measure high-sensitivity CRP and TNF- $\alpha$ , TNF-RI and TNF-R2 (measured at both visits). For exploratory mechanistic analysis, a 10-plex immunoassay of

inflammatory cytokines will be measured at both visits (e.g. IFN- $\gamma$ , IL-1 $\beta$ , IL-2, IL-4, IL-6, IL-8, IL-10, IL-12p70, IL-13). Blood will be collected after a 12 hour fast and centrifuged at 1000g for 15 min at 4°C; plasma will be stored at -80 °C.

*Behavioral assessment:* These tasks are simple, user-friendly tools that provide an opportunity, when used in conjunction with the most widely used questionnaires, to gain novel insights on reward behaviors in mood disorders.

- a) The primary behavioral measurement will be effort-based decision-making, assessed using the Effort-Expenditure for Rewards Task (EEfRT)<sup>33</sup>, which will be done in a fMRI paradigm<sup>73</sup>, as described below during Visits 2 and 3.
- b) Assessments will include the validated anhedonia scale Snaith-Hamilton Pleasure Scale (SHPS), the mood questionnaires Montgomery-Åsberg Depression Rating Scale (MADRS) and Young Mania Rating Scale (YMRS) during each study visit, and the Bandit Task during the first visit.

*Neural Circuits Assessment:* A promising tool to study the effect of insulin on CNS is intranasal insulin, which is delivered directly into the brain, without relevant effects on peripheral glucose<sup>76,77</sup>. A single dose of intranasal insulin has been shown to influence brain activation, increasing regional perfusion and functional connectivity between the hippocampus and the PFC<sup>78-80</sup>. Acute administration of intranasal in randomized, placebo-controlled, cross-over designs has been previously used to determine regional responses to insulin in the resting-state or during tasks<sup>78,80</sup>.

After screening and baseline assessment, participants will receive a crossover treatment assignment of either insulin or diluent followed by an MRI scan, with a washout period of 1 week. Therefore, participants will receive a total of 2 MRI scans throughout the course of the study- one following the first treatment, and one following the second treatment. The subsample will be enriched for the presence of self-reported anhedonia, using a score of greater than 2 on the SHPS as a cut-off, which provides the best discrimination between "normal" and "abnormal" level of hedonic tone<sup>81</sup>. This subsample will also have equal representation of normal weight and obese participants.

To proxy insulin activity within pre-selected brain regions, we will use a provocation paradigm, involving the administration of exogenous intranasal insulin, based on the published work of other research groups<sup>78-80</sup>. Activation of brain regions will be assessed during the resting state and task-based reward paradigm (i.e. EEfRT), following an intranasal administration of either 160 units of intranasal insulin or diluent (insulin and placebo will be prepared as nasal sprays), in a randomized, double-blinded, cross-over design. Please refer to the pharmacy manual for randomization details. A hypothesis-driven region of interest approach will be used to investigate initially the striatum and the medial PFC (mPFC). Willingness to make effort for rewards will be measured with the EEfRT<sup>33</sup>. Briefly, participants have to select between an easy and a hard task. Both tasks involve pressing a key for a predetermined amount of time. The hard task offers more money (variable amounts), but is harder and takes twice as long. Participants make their selection knowingly under different win probabilities (i.e. they might not win money even if they are successful if the win probabilities are low). This task will measure proportions of hard-task choices with varying probabilities of reward and reward magnitudes. To provide stable estimations, the fMRI task will be conducted in three runs<sup>73</sup>.

Table 1

| Assessment | Baseline (V1) | First Spray (V2) | Second Spray (V3) |
|---|---|---|---|
| <b>General Information</b> | | | |
| Demographics | ✓ | | |
| Questionnaire | | | |
| Medical Comorbidity | ✓ | | |
| Questionnaire | | | |
| Family Psychiatric | ✓ | | |
| History | | | |
| Questionnaire | , | | |
| SES Questionnaire | <b>√</b> | | |
| MRI Questionnaire | ✓ | ✓ | ✓ |
| Anthropometric Measures | | | |
| Height (ft) | ✓ | | |
| Weight (kg) | ✓ | ✓ | ✓ |
| Blood Pressure | ✓ | ✓ | ✓ |
| (mmHg) | | | |
| Heart Rate (bpm) | ✓ | ✓ | ✓ |
| Waist/hip | ✓ | | |
| Circumference (cm) | | | |
| Physical Activity/ | ✓ | ✓ | ✓ |
| Energy Expenditure/ | | | |
| 7-Day Accelerometer | | | |
| Wear Time Log | | | |
| Laboratory Assessme | | | |
| Triglycerides | <b>√</b> | <b>√</b> | <b>√</b> |
| Total Cholesterol | <b>√</b> | <b>√</b> | <b>√</b> |
| Insulin | <b>√</b> | <b>√</b> | <b>√</b> |
| Glucose | ✓ | ✓ | ✓ |
| HbA1c | ✓ | ✓ | ✓ |
| C-Peptide | ✓ | ✓ | ✓ |
| IGF-1 | ✓ | ✓ | ✓ |
| TSH | ✓ | ✓ | ✓ |
| Free T4 | ✓ | ✓ | ✓ |
| Free T3 | ✓ | ✓ | ✓ |
| C-Reactive Protein | ✓ | ✓ | ✓ |
| hCG | ✓ | | |
| Imaging | | | |
| fMRI-EEfRT | | ✓ | ✓ |
| Dimensional Measures | | | |
| Clinician Administered | | | |
| YMRS | ✓ | ✓ | ✓ |
| MADRS | ✓ | ✓ | ✓ |
| Bandit Task | ✓ | | |
| Self-Report | | | |

| SHPS | ✓ | ✓ | ✓ |
|----------------------|----------|----------|----------|
| PDQ-D | ✓ | | |
| SDS | ✓ | | |
| UCLA Life Stress | ✓ | | |
| Interview (Episodic) | | | |
| CTQ | ✓ | | |
| DeJong Gierveld | ✓ | | |
| Loneliness Scale | | | |
| Diet History | ✓ | | |
| Questionnaire (III) | | | |
| IPAQ | ✓ | | |
| PSQI | ✓ | | |
| Neurocognitive Tasks | | | |
| DSST | <b>√</b> | <u> </u> | <b>√</b> |
| RAVLT | ✓ | ✓ | ✓ |
| TMT A/B | ✓ | ✓ | ✓ |

Imaging procedures will be started with a safety monitoring for glucose and cardiovascular vital signs. An insulin/placebo spray will be administered intranasally and, within 30 min, fMRI measurement will be performed. Venous blood samples, for determination of plasma glucose and insulin concentrations, will be obtained at the time of the insulin/placebo spray administration and immediately after the scan. The 2 scans for each individuals will be acquired on the same scanner. Subjects will be scanned using a 3.0-Tesla Signa HDx scanner with an 8-channel phased-array receiver coil (GE Healthcare, Milwaukee, Wisconsin) consisting of a structural and functional neuroimaging, comprising:

- Whole-brain 3-D T1-weighted Inversion-Recovery prepared Fast Spoiled Gradient-Echo (IRi. FSPGR) anatomical scan with the following parameters: (TI/TR/TE = 450/8/3 ms, matrix size 256  $\times$  256, field of view 22  $\times$  22 cm, slice thickness = 1 mm, and flip angle = 15°)
- Whole-brain, T2\*-weighted BOLD echo planar imaging (EPI) during awake resting state with the ii. following parameters: (TR/TE = 2000/30 ms, 3.5 x 3.5 x 3.5 mm voxel size, field of view 24x24 cm, 39 slices, slice thickness 3.5 mm, matrix size 64x64, number of frames = 405, flip angle =
- Three runs of whole-brain, T2\*-weighted BOLD EPI series during task-based reward paradigm iii. with the same parameters as in ii.

#### 4. Study Treatment

4.1 Treatments Administered

# Description of Study Medications

The Investigational Pharmacy Services (IPS, also known as the clinical trials pharmacy) at the University Health Network's (UHN's) Toronto Western Hospital (TWH) will be responsible for all study related preparation, dispensing, and documentation. IPS will be responsible for the following study preparation procedures. All active treatment and placebo will be prepared by an IV certified pharmacy technician, under aseptic conditions, in a sterile room, i.e., centralized intravenous additive services (CIVA) area, and verified by a pharmacist.

Dose preparation for the active and placebo nasal sprays follow the same procedure. This will be conducted upon the receipt of an order from the blinded investigator with regard to the number of nasal spray bottles of Humulin® R insulin or diluent to be prepared the pharmacy.

Each product, whether intranasal Humulin<sup>®</sup> R insulin or diluent, will be prepared under the laminar flow hood one at a time. Using aseptic technique, the protective cap is removed from the vial of Humulin® R insulin or diluent (10 mL/vial, manufactured by Eli Lilly) and the rubber stopper is swabbed with an alcohol swab and allowed to dry. Using an appropriate sterile Luer Lock syringe with an appropriately sized needle attached with the bevel of the needle facing up at a 45 degree angle, the Humulin® R insulin or diluent vial is punctured and 5 mL of insulin or diluent is removed and transferred to a metered dose nasal spray bottle (PharmaSystems, Inc.) provided by the study coordinator overseeing the project herein. The nasal spray bottle is then capped accordingly. In summary, the intranasal solutions are prepared as follows:

• Intranasal Insulin Arm: IPS will obtain commercial supplies of Humulin® R insulin (10 mL/vial, manufactured by Eli Lilly) and aseptically transfer a 5 mL sample into a metered dose nasal spray bottle (PharmaSystems Inc.).

Intranasal Placebo Arm: IPS will obtain commercial supplies of Humulin® R insulin's diluent (10 mL/vial, manufactured by Eli Lilly) and aseptically transfer a 5 mL sample into a metered dose nasal spray bottle (PharmaSystems Inc.).

This procedure is repeated until the required number of nasal spray bottles has been prepared. Once completed, the nasal spray bottles are wiped with 70% isopropyl alcohol soaked gauge and removed from the laminar flow hood and appropriately labeled.

Both active and placebo nasal spray bottles are kept separate from each other and a worksheet will be completed to document information, including date of preparation, batch #, expiry date, drug name and strength. The IV certified pharmacy technician who has prepared the dose is responsible for completing the documentation and will be affixing the labels identifying what was prepared. The labels, at a minimum, will contain information regarding the lot #, strength, date of manufacture, expiry date, and storage conditions. All of this will be verified by a pharmacist.

# Labeling

All labels will contain product name, volume, protocol number, investigational drug warning, dosage instructions, storage conditions, lot number, expiration date, and the pharmacy name.

#### **Storage**

Please refer to the pharmacy manual for information on storage.

## **Study Medication Administration**

This will be a single-dose, randomized, double-blinded, cross-over study involving intranasal insulin/placebo solution.

Designated pharmacy staff will dispense study medication, in a double-blind manner, according to the randomization code specific to each subject and dosing period.

Details regarding intranasal insulin and diluent can be referred to in the pharmacy manual.

The investigator and/or designee will instruct the study participant on how the intranasal insulin/placebo spray should be administered. Each study participant is to receive a single dose of Humulin R 160 U / placebo.

- Given:
  - The nasal spray bottles provide a deliverable volume of 0.1 mL/spray.
  - o Humulin R insulin will be sourced as 100 units/mL in a vials of 10 mL from Eli Lilly.
  - o Diluent will be sourced as 10 mL/vial from Eli Lilly.
- Each spray will offer:
  - o 0.1 mL (i.e., 10 units) of Humulin R insulin
  - o 0.1 mL of diluent (to serve as placebo)
- To obtain a dose Humulin R 160 U / placebo
  - o 16 sprays (0.1 mL/spray) are to be given per dose

- o This works out to 16 sprays split between each nostril such that each nostril receives 8 sprays.
- The sprays will be administered between alternating nostrils.

Given this is a crossover study, the study participants will receive a total of two doses in this study. The time between 2 doses is one week.

# 4.2 Accountability of Study Supplies

Please refer to the pharmacy manual for information on accountability of study supplies.

4.3 Disposition of Used/Unused Product

Please refer to the pharmacy manual for information on the disposition of used/unused product.

# 5. Methods of Assigning Subjects to Treatment Groups

Please refer to the pharmacy manual for information on the methods of assigning subjects to treatment groups (i.e. randomization, and blinking/masking).

#### 6. Analytic Plan, Power Analysis and Approach to Potential Challenges

Initial data analyses will inspect socio-demographic and clinical group differences as well as correlations between clinical and biological variables and specified behavioral measures. Clinical or demographic variables demonstrating a correlation with both biological and behavioral measures, will be assessed as potential confounders<sup>82</sup>. The EEfRT behavioral data will be analyzed using generalized estimating equation (GEE) models, according to previous studies<sup>30,33</sup>. For the assessment of associations between the remaining behavioral measurements and biometric data, we will use generalized linear models, due to its greater flexibility and ability to analyze data with non-normal distributions. Group (mood disorders vs. non-psychiatric) effects will be analyzed, with age, gender, and other relevant covariates included in the models. Special considerations will be given to smoking and use psychotropic medications, given its potential effects of both reward processes and insulin signaling.

Mediation and moderation models will be assessed using regression-based, bias-corrected bootstrap tests<sup>83</sup>. The main objective is to test whether there is a mediated effect of X (i.e. mood disorders) on the outcome Y (i.e. anhedonia and reward behavior) through M (i.e. insulin signaling and dopamine metabolism). If appropriate, moderated mediation models (conditional process analysis) will be used to test whether the mediation effect was contingent on a moderating variable W (e.g. obesity, medications). This method uses bootstrapping to determine bias-corrected (asymmetric) 95% confidence intervals for the indirect effects<sup>84</sup>. Bootstrapping methods have been recently advocated, as they are based on random sampling of the data and do not make assumptions about the shape of the sampling distribution; they are also more powerful and allow for the construction of more accurate confidence intervals, relative to normal theory methods<sup>83</sup>.

For the imaging analysis, statistical parametric mapping (SPM8, Wellcome Department of Cognitive Neurology, London, U.K., www.fil.ion.ucl.ac.uk/spm) will be used to preprocess the raw fMRI data. A hypothesis-driven region of interest approach will be used to investigate initially the striatum and mPFC. For the resting-state data, BOLD signal in these regions will be compared between conditions (i.e. insulin and placebo) for each subject using GEE. For the task-based data, mean percent BOLD signal change in these regions under varying reward and probability conditions will be extracted, and we will compute a set of contrasts testing the main effects of reward magnitude, reward

probability, and the interaction for each subject<sup>73</sup>. These first-level individual contrast maps will be fed into a second-level group (i.e. mood disorders vs. controls) and condition analysis, which will also use GEE. Association between behavioral measurements, biometric data and neuroimaging measurements will be assessed with generalized linear models. The false discovery rate (FDR) method will be used to correct for multiple comparisons and significance will be taken at a FDR-corrected threshold of p <  $0.05^{86}$ .

Power Analysis: The primary hypothesis of this study is that anhedonic symptoms in individuals with mood disorders will be mediated by abnormalities in insulin signaling; therefore, the power analysis is based on a bias-corrected bootstrap test of mediation. Results from our preliminary data indicated that the path coefficients were mostly of medium effect sizes (e.g.  $\beta \approx 0.25$ -0.35); empirical analysis indicated that in this condition a sample sizes of 116 is necessary to achieve 80% power85. To account for the possibility of subject attrition and/or inadequate measurements, we will set an initial enrollment goal of 150 subjects.

Potential Challenges and Ways to Overcome Them: The primary challenge in this study is that of recruiting and retaining 150 participants over a 3-year period. Given the experience and volume of the mood disorders clinics involved in this study, we believe that this goal is attainable. There are two potential limitations in our sample composition proposal. First, it is expected that the majority of participants recruited in tertiary mood disorders clinics will report clinically significant anhedonic symptoms. Nonetheless, it is possible that some of the subconstructs analyzed will not display satisfactory psychometric properties for contrast/comparisons. Second, we propose to pre-stratify our sample based on overweight/obesity. There is a well-documented association between adiposity and insulin sensitivity; though these are not perfectly collinear constructs. There are no, however, validated, publicly available, normative data of anhedonic symptoms, whereas gold-standard evaluations of insulin sensitivity are invasive and costly (e.g. hyperinsulinemic euglycemic clamp); therefore approximations are initially necessary. We propose to conduct a preliminary analyses after one third of the sample (n=50) is recruited and reevaluate the sample selection procedures.

A key challenge for the interpretation of results will be how to account for the role of potential confounding factors. These factors include, but are not limited to, psychotropic medications, smoking, socio-demographic characteristics, dietary and lifestyle factors. We opted for a "real-life" naturalistic treatment-seeking sample, as we seek to recruit a sample that is representative of other clinical samples. Moreover, ethical considerations preclude us from withdrawing or deferring initiation of medications. Therefore, we propose to systematically measure these confounding factors and use it as control and/or sub-stratification variables, as appropriate.

#### ADVERSE EVENTS

**Definitions** 

Adverse event

An adverse event is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. An undesirable medical condition can be symptoms (e.g., nausea, chest pain), signs (e.g., tachycardia, enlarged liver) or the abnormal results of an investigation (e.g., laboratory findings, electrocardiogram). In clinical studies, an AE can include an undesirable medical condition occurring at any time, including run-in or washout periods, even if no study treatment has been administered.

#### Serious adverse event

A serious adverse event is an AE occurring during any study phase (i.e., run-in, treatment, washout, follow-up), and at any dose of the investigational product, comparator or placebo, that fulfils one or more of the following criteria:

- results in death
- is immediately life-threatening
- requires in-patient hospitalization or prolongation of existing hospitalization
- results in persistent or significant disability or incapacity
- is a congenital abnormality or birth defect
- is an important medical event that may jeopardize the patient or may require medical intervention to prevent one of the outcomes listed above.

The causality of SAEs (i.e., their relationship to study treatment) will be assessed by the investigator(s). Note that SAEs that could be associated with any study procedure should also be reported. For such events the casual relationship is implied as "yes".

#### Recording of adverse events

AEs will be collected during each visit. At each visit, subjects will be asked if they have had any health problems since the previous visit. All AEs will be recorded appropriately, whether or not considered related to the investigational product. This will include AEs spontaneously reported by the patient and/or observed by the staff as well as AEs reported in response to a direct question e.g. "Have you had any health problems since your last visit?"

For each AE, the following parameters be described:

- start and stop date
- action taken with regards to investigational product
- outcome
- if the AE caused the patient to discontinue
- a statement if the AE fulfils the criteria for a SAE or not
- the investigator's assessment of the causal relationship between the event and the investigational product
  - intensity of the AE
  - o mild (awareness of sign or symptom, but easily tolerated)
  - o moderate (discomfort sufficient to cause interference with normal activities)
  - o severe (incapacitating, with inability to perform normal activities)

It is important to distinguish between serious and severe AEs. Severity is a measure of intensity whereas seriousness is defined by the criteria in Section. An AE of severe intensity need not necessarily be considered serious. For example, nausea that persists for several hours may be considered severe nausea, but not an SAE. On the other hand, a stroke that results in only a limited degree of disability may be considered a mild stroke but would be an SAE.

Symptoms associated with overdose should be reported as AEs. For further information regarding overdose, see section.

Pregnancy in itself is not regarded as an AE unless there is a suspicion that an investigational product may have interfered with the effectiveness of a contraceptive medication.

Follow-up of adverse events should be based upon the clinical judgement of the investigator.

Reporting of serious adverse events

Reporting of SAEs to regulatory authorities will be done by the investigator in accordance with local regulations. A copy of the report will also be sent to the manufacturer of the investigational product.

# 7. Anticipated Timeline

Study start-up is planned immediately after REB approval. The last six months will focus on data management, image processing and analyses. This will allow 27 months of subject recruitment and study execution, with a target of an average of 2-3 participants per site per month.

# 8. Personnel and Facilities

Dr. Rodrigo B. Mansur (co-principal investigator [PI]) is an Assistant Professor of Psychiatry at the University of Toronto and a Clinician-Investigator at the Mood Disorders Psychopharmacology Unit (MDPU) at the University Health Network. His role on the project is to oversee all of the procedures and he will be involved in the design, implementation, and interpretation of all aspects of the study. Dr. Roger S. McIntyre is a Professor of Psychiatry and Pharmacology at the University of Toronto and is Head of MDPU at the University Health Network; he will facilitate the design and implementation of the study and provide clinical and statistical expertise. As clinicians, they will also be involved in subject recruitment and screening. Dr. Jian Chen is the Director of Proteomic Sciences, Indoc Research, and an Assistant Professor at the Department of Pathology and Molecular Medicine, Queen's University. He will be responsible for the proteomic/genomics analysis.

Other Personnel: We will employ part-time research coordinators who will oversee all endeavors related to startup and completion of the study.

Infrastructure and Facilities:

The study will be conducted at the University Health Network (UHN), which is among the largest Health Science Centers in Canada. The investigators will work with a research coordinator, clinicians, and scientists on this project. Investigators all have access to full-service clinical laboratories at UHN. Neuroimaging will be acquired at the Toronto Neuroimaging Facility at the University of Toronto, which has a 3T GE Signa HDx MRI scanners equipped with an 8-channel phased-array head coil.

#### 9. Innovation, Impact and Future Research Plans

The proposed study is the first to integrate an innovative theoretical framework with unique methodological components, which are, nonetheless, extensively supported by the current literature. The study of obesity and insulin sensitivity in mood disorders has often been a secondary concern; this study is among the first to propose approaching metabolic factors as integral to mood disorders pathophysiology. Our proposed methodology includes multiple levels of assessment, using validated tools and techniques, and has the potential to provide a more comprehensive view of insulin's role. We are also proposing a systematic and detailed evaluation of environmental factors, which have a key role on the mood-metabolic disorders comorbidity.

We expect that results from this study will advance the knowledge on the mechanistic basis of anhedonia, which is a critical step for the development of targeted and more effective therapeutic options for individuals with MDD and BD. In addition, by highlighting the role of insulin signaling in the pathophysiology of mood disorders, we hope to refine the conceptual framework on the association between mood and metabolic disorders. Understanding better the impact of insulin signaling disturbances has tremendous potential to reframe how researchers and clinicians conceptualize mood disorders. Ultimately, the aim is to support the development of empirically supported, integrated therapies, such as medications and/or behavioral modifications (e.g. exercise programs) that target both mood and metabolic manifestations. These are urgently necessary to address adequately the multifaceted needs of affected individuals and families.

Future research plans consists of eventually establishing a longitudinal cohort, focused on the interface of metabolic and mood disorders. There is a clear need for longitudinal studies in this area; it is the only design that allows for the exploration of developmental trajectories and for definitive conclusions on causality. Moreover, our research team has ongoing collaborations with international groups, including Brazil, China, Denmark and South Korea, which have generated published articles and collaborative projects; we also intend to further develop these collaborations and explore opportunities for replication studies and cross-cultural comparisons. Finally, our research group has extensive experience with clinical trials, especially with metabolic/inflammatory treatments, such as the immunomodulatory infliximab and the antidiabetic medication liraglutide. We expect that this study will provide opportunities for translational studies, specifically by identifying novel pharmacological targets and/or subgroups of individuals (e.g. obese patients with disturbances in reward valuation) more likely to respond to novel therapies.

#### References

- 1. DALYs GBD, Collaborators H, Murray CJ, Barber RM, Foreman KJ, Ozgoren AA, et al. Global, regional, and national disability-adjusted life years (DALYs) for 306 diseases and injuries and healthy life expectancy (HALE) for 188 countries, 1990-2013: quantifying the epidemiological transition. Lancet. 2015.
- 2. Laursen TM, Musliner KL, Benros ME, Vestergaard M, Munk-Olsen T. Mortality and life expectancy in persons with severe unipolar depression. J Affect Disord. 2016;193:203-7.
- 3. Charlson FJ, Baxter AJ, Dua T, Degenhardt L, Whiteford HA, Vos T. Excess Mortality from Mental, Neurological, and Substance Use Disorders in the Global Burden of Disease Study 2010. In: Patel V, Chisholm D, Dua T, Laxminarayan R, Medina-Mora ME, editors. Mental, Neurological, and Substance Use Disorders: Disease Control Priorities, Third Edition (Volume 4). Washington (DC)2016.
- 4. Nefs G, Pop VJ, Denollet J, Pouwer F. Depressive symptoms and all-cause mortality in people with type 2 diabetes: a focus on potential mechanisms. Br J Psychiatry. 2016;209(2):142-9.
- 5. Nefs G, Pouwer F, Denollet J, Kramer H, Wijnands-van Gent CJ, Pop VJ. Suboptimal glycemic control in type 2 diabetes: a key role for anhedonia? J Psychiatr Res. 2012;46(4):549-54.
- 6. Vancampfort D, Mitchell AJ, De Hert M, Sienaert P, Probst M, Buys R, et al. Type 2 Diabetes in Patients with Major Depressive Disorder: A Meta-Analysis of Prevalence Estimates and Predictors. Depress Anxiety. 2015;32(10):763-73.
- 7. Vancampfort D, Stubbs B, Mitchell AJ, De Hert M, Wampers M, Ward PB, et al. Risk of metabolic syndrome and its components in people with schizophrenia and related psychotic disorders, bipolar disorder and major depressive disorder: a systematic review and meta-analysis. World Psychiatry. 2015;14(3):339-47.
- 8. Luppino FS, de Wit LM, Bouvy PF, Stijnen T, Cuijpers P, Penninx BW, et al. Overweight, obesity, and depression: a systematic review and meta-analysis of longitudinal studies. Arch Gen Psychiatry. 2010;67(3):220-9.
- 9. Pan A, Keum N, Okereke OI, Sun Q, Kivimaki M, Rubin RR, et al. Bidirectional association between depression and metabolic syndrome: a systematic review and meta-analysis of epidemiological studies. Diabetes Care. 2012;35(5):1171-80.
- 10. Mannan M, Mamun A, Doi S, Clavarino A. Is there a bi-directional relationship between depression and obesity among adult men and women? Systematic review and bias-adjusted meta analysis. Asian J Psychiatr. 2016;21:51-66.
- 11. Wahlqvist ML, Lee MS, Chuang SY, Hsu CC, Tsai HN, Yu SH, et al. Increased risk of affective disorders in type 2 diabetes is minimized by sulfonylurea and metformin combination: a population-based cohort study. BMC Med. 2012;10:150.
- 12. Kumar A, Gupta R, Thomas A, Ajilore O, Hellemann G. Focal subcortical biophysical abnormalities in patients diagnosed with type 2 diabetes and depression. Arch Gen Psychiatry. 2009;66(3):324-30.
- 13. Ajilore O, Narr K, Rosenthal J, Pham D, Hamilton L, Watari K, et al. Regional cortical gray matter thickness differences associated with type 2 diabetes and major depression. Psychiatry Res. 2010;184(2):63-70.

- Zhou JX, Li HC, Bai XJ, Chang BC, Li CJ, Sun P, et al. Functional Val66Met polymorphism of Brain-derived neurotrophic factor in type 2 diabetes with depression in Han Chinese subjects. Behav Brain Funct. 2013;9:34.
- 15. Amare AT, Schubert KO, Klingler-Hoffmann M, Cohen-Woods S, Baune BT. The genetic overlap between mood disorders and cardiometabolic diseases: a systematic review of genome wide and candidate gene studies. Transl Psychiatry. 2017;7(1):e1007.
- 16. Covinsky KE, Cenzer IS, Yaffe K, O'Brien S, Blazer DG. Dysphoria and anhedonia as risk factors for disability or death in older persons: implications for the assessment of geriatric depression. Am J Geriatr Psychiatry. 2014;22(6):606-13.
- 17 McMakin DL, Olino TM, Porta G, Dietz LJ, Emslie G, Clarke G, et al. Anhedonia predicts poorer recovery among youth with selective serotonin reuptake inhibitor treatment-resistant depression. J Am Acad Child Adolesc Psychiatry. 2012;51(4):404-11.
- Turner AD, Capuano AW, Wilson RS, Barnes LL. Depressive symptoms and cognitive decline in older african americans: two scales and their factors. Am J Geriatr Psychiatry. 2015;23(6):568-78.
- 19. Vinckier F, Gourion D, Mouchabac S. Anhedonia predicts poor psychosocial functioning: Results from a large cohort of patients treated for major depressive disorder by general practitioners. Eur Psychiatry. 2017;44:1-8.
- McCabe C, Mishor Z, Cowen PJ, Harmer CJ. Diminished neural processing of aversive and 20. rewarding stimuli during selective serotonin reuptake inhibitor treatment. Biol Psychiatry. 2010;67(5):439-45.
- 21. Nierenberg AA, Husain MM, Trivedi MH, Fava M, Warden D, Wisniewski SR, et al. Residual symptoms after remission of major depressive disorder with citalogram and risk of relapse: a STAR\*D report. Psychol Med. 2010;40(1):41-50.
- 22. Nierenberg AA, Keefe BR, Leslie VC, Alpert JE, Pava JA, Worthington JJ, 3rd, et al. Residual symptoms in depressed patients who respond acutely to fluoxetine. J Clin Psychiatry. 1999;60(4):221-5.
- Nusslock R, Alloy LB. Reward processing and mood-related symptoms: An RDoC and 23. translational neuroscience perspective. J Affect Disord. 2017;216:3-16.
- Rizvi SJ, Pizzagalli DA, Sproule BA, Kennedy SH. Assessing anhedonia in depression: 24. Potentials and pitfalls. Neurosci Biobehav Rev. 2016;65:21-35.
- Thomsen KR. Measuring anhedonia: impaired ability to pursue, experience, and learn about reward. Front Psychol. 2015;6:1409.
- 26. Kozak MJ, Cuthbert BN. The NIMH Research Domain Criteria Initiative: Background, Issues, and Pragmatics. Psychophysiology. 2016;53(3):286-97.
- 27. Criteria NAMHCWoTaMfRD. Behavioral Assessment Methods for RDoC Constructs. . Bethesda, MD.: 2016.
- 28. Sherdell L, Waugh CE, Gotlib IH. Anticipatory pleasure predicts motivation for reward in major depression. J Abnorm Psychol. 2012;121(1):51-60.

- Treadway MT, Bossaller NA, Shelton RC, Zald DH. Effort-based decision-making in major depressive disorder: a translational model of motivational anhedonia. J Abnorm Psychol. 2012;121(3):553-8.
- 30. Yang XH, Huang J, Zhu CY, Wang YF, Cheung EF, Chan RC, et al. Motivational deficits in effort-based decision making in individuals with subsyndromal depression, first-episode and remitted depression patients. Psychiatry Res. 2014;220(3):874-82.
- 31. Clery-Melin ML, Schmidt L, Lafargue G, Baup N, Fossati P, Pessiglione M. Why don't you try harder? An investigation of effort production in major depression. PLoS One. 2011;6(8):e23178.
- 32. Pizzagalli DA, Jahn AL, O'Shea JP. Toward an objective characterization of an anhedonic phenotype: a signal-detection approach. Biol Psychiatry. 2005;57(4):319-27.
- 33. Treadway MT, Buckholtz JW, Schwartzman AN, Lambert WE, Zald DH. Worth the 'EEfRT'? The effort expenditure for rewards task as an objective measure of motivation and anhedonia. PLoS One. 2009;4(8):e6598.
- 34. Russo SJ, Nestler EJ. The brain reward circuitry in mood disorders. Nat Rev Neurosci. 2013;14(9):609-25.
- 35. Haber SN, Knutson B. The reward circuit: linking primate anatomy and human imaging. Neuropsychopharmacology. 2010;35(1):4-26.
- Ballard IC, Murty VP, Carter RM, MacInnes JJ, Huettel SA, Adcock RA. Dorsolateral 36. prefrontal cortex drives mesolimbic dopaminergic regions to initiate motivated behavior. J Neurosci. 2011;31(28):10340-6.
- 37. Young CB, Chen T, Nusslock R, Keller J, Schatzberg AF, Menon V. Anhedonia and general distress show dissociable ventromedial prefrontal cortex connectivity in major depressive disorder. Transl Psychiatry. 2016;6:e810.
- 38. Zhang B, Lin P, Shi H, Ongur D, Auerbach RP, Wang X, et al. Mapping anhedonia-specific dysfunction in a transdiagnostic approach: an ALE meta-analysis. Brain Imaging Behav. 2016;10(3):920-39.
- Berridge KC, Robinson TE. What is the role of dopamine in reward: hedonic impact, reward learning, or incentive salience? Brain Res Brain Res Rev. 1998;28(3):309-69.
- 40. Beierholm U, Guitart-Masip M, Economides M, Chowdhury R, Duzel E, Dolan R, et al. Dopamine modulates reward-related vigor. Neuropsychopharmacology. 2013;38(8):1495-503.
- 41. Steinberg EE, Keiflin R, Boivin JR, Witten IB, Deisseroth K, Janak PH. A causal link between prediction errors, dopamine neurons and learning. Nat Neurosci. 2013;16(7):966-73.
- Hamid AA, Pettibone JR, Mabrouk OS, Hetrick VL, Schmidt R, Vander Weele CM, et al. Mesolimbic dopamine signals the value of work. Nat Neurosci. 2016;19(1):117-26.
- Sarchiapone M, Carli V, Camardese G, Cuomo C, Di Giuda D, Calcagni ML, et al. Dopamine 43 transporter binding in depressed patients with anhedonia. Psychiatry Res. 2006;147(2-3):243-8.

- Cannon DM, Klaver JM, Peck SA, Rallis-Voak D, Erickson K, Drevets WC. Dopamine type-1 receptor binding in major depressive disorder assessed using positron emission tomography and [11C]NNC-112. Neuropsychopharmacology. 2009;34(5):1277-87.
- 45. Camardese G, De Risio L, Di Nicola M, Pucci L, Cocciolillo F, Bria P, et al. Changes of dopamine transporter availability in depressed patients with and without anhedonia: a 123I-N-omegafluoropropyl-carbomethoxy-3beta- (4-Iodophenyl)tropane SPECT study. Neuropsychobiology. 2014;70(4):235-43.
- Docherty AR, Sponheim SR. Anhedonia as a phenotype for the Val158Met COMT 46. polymorphism in relatives of patients with schizophrenia. J Abnorm Psychol. 2008;117(4):788-98.
- 47 Ceaser A, Csernansky JG, Barch DM. COMT influences on prefrontal and striatal blood oxygenation level-dependent responses during working memory among individuals with schizophrenia, their siblings, and healthy controls. Cogn Neuropsychiatry. 2013;18(4):257-83.
- 48. Bogdan R, Nikolova YS, Pizzagalli DA. Neurogenetics of depression: a focus on reward processing and stress sensitivity. Neurobiol Dis. 2013;52:12-23.
- 49. Figlewicz DP, Sipols AJ. Energy regulatory signals and food reward. Pharmacol Biochem Behav. 2010;97(1):15-24.
- 50. Shaw LM. The insulin receptor substrate (IRS) proteins: at the intersection of metabolism and cancer. Cell Cycle. 2011;10(11):1750-6.
- 51. White MF. Regulating insulin signaling and beta-cell function through IRS proteins. Can J Physiol Pharmacol. 2006;84(7):725-37.
- Lin X, Taguchi A, Park S, Kushner JA, Li F, Li Y, et al. Dysregulation of insulin receptor substrate 2 in beta cells and brain causes obesity and diabetes. J Clin Invest. 2004:114(7):908-16.
- 53. Pardini AW, Nguyen HT, Figlewicz DP, Baskin DG, Williams DL, Kim F, et al. Distribution of insulin receptor substrate-2 in brain areas involved in energy homeostasis. Brain Res. 2006;1112(1):169-78.
- Costello DA, Claret M, Al-Qassab H, Plattner F, Irvine EE, Choudhury AI, et al. Brain deletion of insulin receptor substrate 2 disrupts hippocampal synaptic plasticity and metaplasticity. PLoS One. 2012;7(2):e31124.
- 55. Heni M, Kullmann S, Preissl H, Fritsche A, Haring HU. Impaired insulin action in the human brain: causes and metabolic consequences. Nat Rev Endocrinol, 2015;11(12):701-11.
- 56. Biessels GJ, Reagan LP. Hippocampal insulin resistance and cognitive dysfunction. Nat Rev Neurosci. 2015;16(11):660-71.
- 57. Kullmann S, Heni M, Fritsche A, Preissl H. Insulin action in the human brain: evidence from neuroimaging studies. J Neuroendocrinol. 2015;27(6):419-23.
- Beeler JA, Frazier CR, Zhuang X. Putting desire on a budget: dopamine and energy expenditure, reconciling reward and resources. Front Integr Neurosci. 2012;6:49.

- 59. Khanh DV, Choi YH, Moh SH, Kinyua AW, Kim KW. Leptin and insulin signaling in dopaminergic neurons: relationship between energy balance and reward system. Front Psychol. 2014;5:846.
- 60. Bradberry CW, Karasic DH, Deutch AY, Roth RH. Regionally-specific alterations in mesotelencephalic dopamine synthesis in diabetic rats: association with precursor tyrosine. J Neural Transm Gen Sect. 1989;78(3):221-9.
- 61. Kono T, Takada M. Dopamine depletion in nigrostriatal neurons in the genetically diabetic rat. Brain Res. 1994;634(1):155-8.
- 62. Dunn JP, Kessler RM, Feurer ID, Volkow ND, Patterson BW, Ansari MS, et al. Relationship of dopamine type 2 receptor binding potential with fasting neuroendocrine hormones and insulin sensitivity in human obesity. Diabetes Care. 2012;35(5):1105-11.
- 63. Caravaggio F, Borlido C, Hahn M, Feng Z, Fervaha G, Gerretsen P, et al. Reduced insulin sensitivity is related to less endogenous dopamine at D2/3 receptors in the ventral striatum of healthy nonobese humans. Int J Neuropsychopharmacol. 2015;18(7):pyv014.
- 64. Steele KE, Prokopowicz GP, Schweitzer MA, Magunsuon TH, Lidor AO, Kuwabawa H, et al. Alterations of central dopamine receptors before and after gastric bypass surgery. Obes Surg. 2010;20(3):369-74.
- 65. Figlewicz DP, Brot MD, McCall AL, Szot P. Diabetes causes differential changes in CNS noradrenergic and dopaminergic neurons in the rat: a molecular study. Brain Res. 1996;736(1-2):54-60.
- 66. Petrisic MS, Augood SJ, Bicknell RJ. Monoamine transporter gene expression in the central nervous system in diabetes mellitus. J Neurochem. 1997;68(6):2435-41.
- 67. Wang JP, Liu IM, Tzeng TF, Cheng JT. Decrease in catechol-O-methyltransferase activity in the liver of streptozotocin-induced diabetic rats. Clin Exp Pharmacol Physiol. 2002;29(5-6):419-22.
- 68. Kleinridders A, Cai W, Cappellucci L, Ghazarian A, Collins WR, Vienberg SG, et al. Insulin resistance in brain alters dopamine turnover and causes behavioral disorders. Proc Natl Acad Sci U S A. 2015;112(11):3463-8.
- 69. Eisenstein SA, Gredysa DM, Antenor-Dorsey JA, Green L, Arbelaez AM, Koller JM, et al. Insulin, Central Dopamine D2 Receptors, and Monetary Reward Discounting in Obesity. PLoS One. 2015;10(7):e0133621.
- 70. Xu N, Geller DH, Jones MR, Funari VA, Azziz R, Goodarzi MO. Comprehensive assessment of expression of insulin signaling pathway components in subcutaneous adipose tissue of women with and without polycystic ovary syndrome. J Clin Transl Endocrinol. 2015;2(3):99-104.
- 71. Blum K, Thanos PK, Gold MS. Dopamine and glucose, obesity, and reward deficiency syndrome. Front Psychol. 2014;5:919.
- 72. Purves-Tyson TD, Owens SJ, Rothmond DA, Halliday GM, Double KL, Stevens J, et al. Putative presynaptic dopamine dysregulation in schizophrenia is supported by molecular evidence from post-mortem human midbrain. Transl Psychiatry. 2017;7(1):e1003.

- Yang XH, Huang J, Lan Y, Zhu CY, Liu XQ, Wang YF, et al. Diminished caudate and superior temporal gyrus responses to effort-based decision making in patients with first-episode major depressive disorder. Prog Neuropsychopharmacol Biol Psychiatry. 2016;64:52-9.
- 74. Knutson B, Heinz A. Probing psychiatric symptoms with the monetary incentive delay task. Biol Psychiatry. 2015;77(5):418-20.
- Levy I, Snell J, Nelson AJ, Rustichini A, Glimcher PW. Neural representation of subjective 75. value under risk and ambiguity. J Neurophysiol. 2010;103(2):1036-47.
- Kern W, Born J, Schreiber H, Fehm HL. Central nervous system effects of intranasally administered insulin during euglycemia in men. Diabetes. 1999;48(3):557-63.
- Ott V, Benedict C, Schultes B, Born J, Hallschmid M. Intranasal administration of insulin to the brain impacts cognitive function and peripheral metabolism. Diabetes Obes Metab. 2012;14(3):214-21.
- 78. Kullmann S, Heni M, Veit R, Scheffler K, Machann J, Haring HU, et al. Selective insulin resistance in homeostatic and cognitive control brain areas in overweight and obese adults. Diabetes Care. 2015;38(6):1044-50.
- Kullmann S, Frank S, Heni M, Ketterer C, Veit R, Haring HU, et al. Intranasal insulin modulates intrinsic reward and prefrontal circuitry of the human brain in lean women. Neuroendocrinology. 2013;97(2):176-82.
- 80. Zhang H, Hao Y, Manor B, Novak P, Milberg W, Zhang J, et al. Intranasal insulin enhanced resting-state functional connectivity of hippocampal regions in type 2 diabetes. Diabetes. 2015;64(3):1025-34.
- 81. Snaith RP, Hamilton M, Morley S, Humayan A, Hargreaves D, Trigwell P. A scale for the assessment of hedonic tone the Snaith-Hamilton Pleasure Scale. Br J Psychiatry, 1995:167(1):99-103.
- 82. Assmann SF, Pocock SJ, Enos LE, Kasten LE. Subgroup analysis and other (mis)uses of baseline data in clinical trials. Lancet. 2000;355(9209):1064-9.
- 83. Hayes AF. Introduction to Mediation, Moderation, and Conditional Process Analysis: A Regression-Based Approach. New York: Guilford Press; 2013.
- Preacher KJ, Hayes AF. Asymptotic and resampling strategies for assessing and comparing 84. indirect effects in multiple mediator models. Behav Res Methods. 2008;40(3):879-91.
- Fritz MS, Mackinnon DP. Required sample size to detect the mediated effect. Psychol Sci. 85. 2007;18(3):233-9.
- Benjamini Y, Hochberg Y. Controlling the False Discovery Rate: A Practical and Powerful 86. Approach to Multiple Testing Journal of the Royal Statistical Society Series B (Methodological). 1995;57(1):289-300.